CLINICAL TRIAL: NCT00242580
Title: A 24-month Randomized, Double-masked, Sham Controlled, Multicenter, Phase IIIB Study Comparing Photodynamic Therapy With Verteporfin (Visudyne®) Plus Two Different Dose Regimens of Intravitreal Triamcinolone Acetonide (1 mg and 4 mg) Versus Visudyne® Plus Intravitreal Pegaptanib(Macugen®) in Patients With Subfoveal Choroidal Neovascularization Secondary to Age-related Macular Degeneration
Brief Title: A Safety and Efficacy Study Comparing the Combination Treatments of Verteporfin Therapy Plus One of Two Different Doses of Intravitreal Triamcinolone Acetonide and the Verteporfin Therapy Plus Intravitreal Pegaptanib
Acronym: VERITAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: QLT Inc. (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBPD952E2202
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Results first posted 2011-05-02 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Macular Degeneration; Choroidal Neovascularization
Keywords: AMD; age-related macular degeneration; choroidal neovascularization
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Verteporfin; pegaptanib; Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Verteporfin and Triamcinolone 1 mg (Experimental): Participants received Verteporfin photodynamic therapy and 1 mg triamcinolone acetonide intravitreal injection at the baseline visit. After the baseline visit, these participants received Verteporfin and triamcinolone acetonide 1 mg at every 3 month visit up to Month 9 only if leakage was detected on the fluorescein angiogram. At the 1.5, 4.5, 7.5 and 10.5 month follow-up visits participants received a sham injection. Starting from Month 12, if patients experienced ≥ 10 letters vision loss from the previous visit, they were treated at the investigators' discretion with available standard of care therapy.
  Interventions: Drug: Verteporfin photodynamic therapy; Drug: Triamcinolone acetonide
- Verteporfin and Triamcinolone 4 mg (Experimental): Participants received Verteporfin photodynamic therapy and 4 mg triamcinolone acetonide intravitreal injection at the baseline visit. After the baseline visit, these participants received Verteporfin and triamcinolone acetonide 4 mg at every 3 month visit up to Month 9 only if leakage was detected on the fluorescein angiogram. At the 1.5, 4.5, 7.5 and 10.5 month follow-up visits participants received a sham injection. Starting from Month 12, if patients experienced ≥ 10 letters vision loss from the previous visit, they were treated at the investigators' discretion with available standard of care therapy.
  Interventions: Drug: Verteporfin photodynamic therapy; Drug: Triamcinolone acetonide
- Verteporfin and Pegaptanib (Active Comparator): Participants received Verteporfin photodynamic therapy and 0.3 mg Pegaptanib at the baseline visit. After the baseline visit, these participants received pegaptanib every 1.5 months up until and including the 10.5 month visit. After the baseline visit, these participants also received verteporfin at every 3 month visit up to Month 9 only if leakage was detected on the fluorescein angiogram. Starting from Month 12, if participants experienced ≥ 10 letters vision loss from the previous visit, they were treated at the investigator's discretion with available standard of care therapy.
  Interventions: Drug: Verteporfin photodynamic therapy; Drug: Pegaptanib

INTERVENTIONS:
Drug: Verteporfin photodynamic therapy — After a 10-minute intravenous infusion of verteporfin at a dose of 6 mg/m^2 body surface area, verteporfin was activated by light application of 50 J/cm^2 to the study eye, begun 15 minutes after the start of infusion.
  Other Names: Visudyne
Drug: Pegaptanib — Pegaptanib sodium 0.3 mg administered by intravitreal injection.
  Other Names: Macugen
  Arms: Verteporfin and Pegaptanib
Drug: Triamcinolone acetonide — Triamcinolone acetonide administered by intravitreal injection.
  Other Names: Kenalog-40®
  Arms: Verteporfin and Triamcinolone 1 mg; Verteporfin and Triamcinolone 4 mg

SUMMARY:
To evaluate the safety and efficacy of the combination treatments in wet age-related macular degeneration. The combination treatment consists of verteporfin photodynamic therapy and either triamcinolone acetonide or pegaptanib added as an intravitreal injection.

ELIGIBILITY:
Inclusion Criteria:

* age >50
* all types of untreated subfoveal choroidal neovascularization secondary to AMD
* lesion size <5400 microns in greater linear dimension (GLD)

Exclusion Criteria:

* have a history of prior photodynamic therapy, external beam radiation, subfoveal focal laser photocoagulation, submacular surgery, or transpupillary thermotherapy
* known allergy to verteporfin, triamcinolone or pegaptanib
* have received prior treatment with Macugen, or other anti-angiogenic compound or any investigational treatment (e.g. Ruboxistaurin, Lucentis [ranibizumab], Retaane [anecortave acetate], squalamine, siRNA, VEGF-Trap etc.) for neovascular AMD
* have the presence of fibrosis, hemorrhage, pigment epithelial detachments, tear (tip) of the retinal pigment epithelium or other hypoflourescent lesions obscuring greater than 50% of the CNV lesion
* have had previous pars plana vitrectomy in the study eye

Other protocol-specified inclusion/exclusion criteria applied.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2005-09; Primary Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigational Site, Austin, Texas, United States

REFERENCES:
- See also: Novartis patient recruitment website: Clinical trial information for patients and caregivers — http://www.novartisclinicaltrials.com/etrials/DiseaseID83/Age-Related-Macular-Degeneration-clinical-trials.go

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol was amended to limit the sample size from 339 to 100. 111 entered the study and and were part of the 12 mo analysis. The study was subsequently terminated. The patients did not receive study drug during the second year of the study.
Groups:
- Verteporfin + 1 mg Triamcinolone: Participants received Verteporfin photodynamic therapy and 1 mg triamcinolone acetonide intravitreal injection at the baseline visit. After the baseline visit, these participants received Verteporfin and triamcinolone acetonide 1 mg at every 3 month visit up to Month 9 only if leakage was detected on the fluorescein angiogram. At the 1.5, 4.5, 7.5 and 10.5 month follow-up visits participants received a sham injection. Starting from Month 12, if patients experienced ≥ 10 letters vision loss from the previous visit, they were treated at the investigators' discretion with available standard of care therapy.
- Verteporfin + 4 mg Triamcinolone: Participants received Verteporfin photodynamic therapy and 4 mg triamcinolone acetonide intravitreal injection at the baseline visit. After the baseline visit, these participants received Verteporfin and triamcinolone acetonide 4 mg at every 3 month visit up to Month 9 only if leakage was detected on the fluorescein angiogram. At the 1.5, 4.5, 7.5 and 10.5 month follow-up visits participants received a sham injection. Starting from Month 12, if patients experienced ≥ 10 letters vision loss from the previous visit, they were treated at the investigators' discretion with available standard of care therapy.
- Verteporfin + Pegaptanib: Participants received Verteporfin photodynamic therapy and 0.3 mg Pegaptanib at the baseline visit. After the baseline visit, these participants received pegaptanib every 1.5 months up until and including the 10.5 month visit. After the baseline visit, these participants also received verteporfin at every 3 month visit up to Month 9 only if leakage was detected on the fluorescein angiogram. Starting from Month 12, if participants experienced ≥ 10 letters vision loss from the previous visit, they were treated at the investigator's discretion with available standard of care therapy.
Period: Overall Study
Arm/Group | Verteporfin + 1 mg Triamcinolone | Verteporfin + 4 mg Triamcinolone | Verteporfin + Pegaptanib
Started | 32 | 41 | 38
Completed | 22 ("Completed" indicates 12 month data.) | 29 | 24
Not Completed | 10 | 12 | 14
Not completed — Adverse Event | 3 | 0 | 2
Not completed — Unsatisfactory therapeutic effect | 4 | 5 | 5
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Subject withdrew consent | 2 | 2 | 5
Not completed — Lost to Follow-up | 0 | 3 | 0
Not completed — Death | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Verteporfin + 1 mg Triamcinolone | Verteporfin + 4 mg Triamcinolone | Verteporfin + Pegaptanib | Total
Number analyzed (Participants) | 32 | 41 | 38 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (9) | 78 (8) | 81 (6) | 78 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 25 | 20 | 63
  Male | 14 | 16 | 18 | 48
Region of Enrollment [Number; unit: participants]
  United States | 32 | 41 | 38 | 111

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Lose Less Than 15 Letters of Best Corrected Visual Acuity (BCVA) at 12 Months From Baseline.
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An ETDRS visual acuity score of 85 is approximately 20/20. A decrease in score indicates worsening of vision. This outcome assessed the percentage of participants who lost less than 15 letters of visual acuity at 12 months as compared with baseline.
Time Frame: Baseline to Month 12
Population: Intent-to-treat (ITT) data set includes data from all randomized patients. Missing data were imputed using last observation carried forward.
Measure: Number; unit: Percentage of Participants
Arm/Group | Verteporfin + 1 mg Triamcinolone | Verteporfin + 4 mg Triamcinolone | Verteporfin + Pegaptanib
Number analyzed (Participants) | 32 | 41 | 38
Percentage of Participants | 59.4 | 63.4 | 71.1

2. Secondary Outcome: Percentage of Participants With Gain of 5 or More Letters of Best Corrected Visual Acuity From Baseline to Month 12
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An ETDRS visual acuity score of 85 is approximately 20/20. An increased score indicates improvement in acuity. This outcome assessed the percentage of participants who gained 5 or more letters of visual acuity at 12 months compared with baseline.
Time Frame: Baseline to Month 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Verteporfin + 1 mg Triamcinolone | Verteporfin + 4 mg Triamcinolone | Verteporfin + Pegaptanib
Number analyzed (Participants) | 32 | 41 | 38
Percentage of Participants | 31.3 | 12.2 | 28.9

3. Secondary Outcome: Percentage of Participants With Gain of BCVA of 10 or More Letters at 12 Months
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An ETDRS visual acuity score of 85 is approximately 20/20. An increased score indicates improvement in acuity. This outcome assessed the percentage of participants who gained 10 or more letters of visual acuity at 12 months as compared with baseline.
Time Frame: Baseline to Month 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Verteporfin + 1 mg Triamcinolone | Verteporfin + 4 mg Triamcinolone | Verteporfin + Pegaptanib
Number analyzed (Participants) | 32 | 41 | 38
Percentage of Participants | 18.8 | 2.4 | 23.7

4. Secondary Outcome: Percentage of Participants With Gain of BCVA Score of 15 or More Letters at Month 12
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An ETDRS visual acuity score of 85 is approximately 20/20. An increased score indicates improvement in acuity. This outcome assessed the percentage of participants who gained 15 or more letters of visual acuity at 12 months as compared with baseline.
Time Frame: Baseline to Month 12
Population: Efficacy variable analyses were performed on the intent-to-treat (ITT) data set. The ITT set includes data from all randomized patients. Missing data were imputed using last observation carried forward.
Measure: Number; unit: Percentage of Participants
Arm/Group | Verteporfin + 1 mg Triamcinolone | Verteporfin + 4 mg Triamcinolone | Verteporfin + Pegaptanib
Number analyzed (Participants) | 32 | 41 | 38
Percentage of Participants | 6.3 | 0 | 13.2

5. Secondary Outcome: Number of Participants Requiring Verteporfin Treatment Throughout the Study
Description: Participants received study drug at the Baseline visit and subsequent retreatment at 3 month intervals if leakage was detected on the fluorescein angiogram. The cumulative distribution of the number of treatments is shown per arm.
Time Frame: Baseline to Month 12
Population: Observed data.
Measure: Number; unit: Participants
Arm/Group | Verteporfin + 1 mg Triamcinolone | Verteporfin + 4 mg Triamcinolone | Verteporfin + Pegaptanib
Number analyzed (Participants) | 32 | 41 | 38
Participants
  Participants who received 1 treatment | 11 (0) | 12 (0) | 10 (0)
  Participants who received 2 treatments | 10 | 15 | 19
  Participants who received 3 treatments | 9 | 12 | 5
  Participants who received 4 treatments | 2 | 2 | 4

6. Secondary Outcome: Mean Change From Baseline in Total Area of Lesion at 12 Months
Description: Fluorescein angiography (FA) was used to assess total lesion area. All angiographs were sent to the Central Reading Center (CRC) for analysis.
Time Frame: Baseline to Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Verteporfin + 1 mg Triamcinolone | Verteporfin + 4 mg Triamcinolone | Verteporfin + Pegaptanib
Number analyzed (Participants) | 32 | 41 | 38
mm^2
  Baseline | 6.9178 (5.9455) | 5.6400 (3.7154) | 6.3011 (5.4794)
  12 Months | 6.8959 (7.6848) | 5.8149 (4.6465) | 8.6245 (7.1242)
  Change from Baseline | -0.0219 (7.7026) | 0.1749 (4.2357) | 2.3234 (5.9370)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Verteporfin + 1 mg Triamcinolone | Verteporfin + 4 mg Triamcinolone | Verteporfin + Pegaptanib
Serious Adverse Events (participants affected / at risk) | 11/32 | 9/41 | 10/38
Other Adverse Events (participants affected / at risk) | 32/32 | 38/41 | 30/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Verteporfin + 1 mg Triamcinolone (N=32) | Verteporfin + 4 mg Triamcinolone (N=41) | Verteporfin + Pegaptanib (N=38)
ACCIDENTAL INJURY (Injury, poisoning and procedural complications) | 2 | 1 | 3
ANAPHYLACTOID REACTION (Immune system disorders) | 1 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 1
CYST (General disorders) | 0 | 0 | 1
HERNIA (General disorders) | 0 | 1 | 0
INFECTION (Infections and infestations) | 1 | 0 | 0
NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
AORTIC STENOSIS (Vascular disorders) | 0 | 1 | 0
ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 1
ARTERIAL ANOMALY (Vascular disorders) | 0 | 0 | 1
ARTERIAL THROMBOSIS (Vascular disorders) | 1 | 0 | 0
ARTERIOSCLEROSIS (Vascular disorders) | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 0
CONGESTIVE HEART FAILURE (Cardiac disorders) | 1 | 0 | 0
CORONARY ARTERY DISORDER (Cardiac disorders) | 0 | 2 | 1
DEEP THROMBOPHLEBITIS (Vascular disorders) | 0 | 0 | 1
HEART BLOCK (Cardiac disorders) | 1 | 0 | 0
MYOCARDIAL INFARCT (Cardiac disorders) | 0 | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 1 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 | 0 | 2
GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 0 | 0 | 1
PEPTIC ULCER HEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
CEREBRAL INFARCT (Nervous system disorders) | 0 | 2 | 0
CEREBRAL ISCHEMIA (Nervous system disorders) | 1 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1 | 0
ENCEPHALOPATHY (Nervous system disorders) | 0 | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 1
LUNG EDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 2 | 2
ACUTE KIDNEY FAILURE (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Verteporfin + 1 mg Triamcinolone (N=32) | Verteporfin + 4 mg Triamcinolone (N=41) | Verteporfin + Pegaptanib (N=38)
ACCIDENTAL INJURY (Injury, poisoning and procedural complications) | 0 | 2 | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
HEADACHE (Nervous system disorders) | 4 | 1 | 3
INFECTION (Infections and infestations) | 5 | 2 | 0
INJECTION SITE EXTRAVASATION (Injury, poisoning and procedural complications) | 2 | 0 | 3
PAIN (General disorders) | 5 | 4 | 3
CORONARY ARTERY DISORDER (Cardiac disorders) | 0 | 3 | 1
HYPERTENSION (Vascular disorders) | 7 | 7 | 2
DIARRHEA (Gastrointestinal disorders) | 1 | 2 | 2
DYSPEPSIA (Gastrointestinal disorders) | 2 | 2 | 1
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 | 4 | 3
NAUSEA (Gastrointestinal disorders) | 4 | 0 | 3
RECTAL DISORDER (Gastrointestinal disorders) | 0 | 3 | 0
ANEMIA (Blood and lymphatic system disorders) | 0 | 3 | 1
HYPERLIPEMIA (Metabolism and nutrition disorders) | 2 | 0 | 2
PERIPHERAL EDEMA (General disorders) | 2 | 0 | 2
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
ANXIETY (Psychiatric disorders) | 0 | 1 | 2
DEMENTIA (Psychiatric disorders) | 0 | 2 | 2
INSOMNIA (Psychiatric disorders) | 0 | 0 | 3
BRONCHITIS (Infections and infestations) | 2 | 0 | 1
COUGH INCREASED (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
PNEUMONIA (Infections and infestations) | 0 | 1 | 2
RHINITIS (Infections and infestations) | 3 | 6 | 2
SINUSITIS (Infections and infestations) | 2 | 2 | 1
CONTACT DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
AMD PROGRESSION (Fellow eye) (Eye disorders) | 5 | 6 | 7
BLEPHARITIS (Fellow eye) (Eye disorders) | 0 | 0 | 2
CATARACT (Fellow eye) (Eye disorders) | 3 | 4 | 2
CONJUNCTIVITIS (Fellow eye) (Eye disorders) | 2 | 0 | 2
DRY EYES (Fellow eye) (Eye disorders) | 1 | 1 | 4
EYE DISORDER (Fellow eye) (Eye disorders) | 0 | 1 | 2
EYE ITCHING (Fellow eye) (Eye disorders) | 2 | 0 | 0
RETINAL DISORDER (Fellow eye) (Eye disorders) | 2 | 3 | 2
RETINAL HEMORRHAGE (Fellow eye) (Eye disorders) | 1 | 0 | 2
SUBRETINAL HEMORRHAGE (Fellow eye) (Eye disorders) | 2 | 0 | 0
TINNITUS (Ear and labyrinth disorders) | 0 | 0 | 2
VISION DECREASED (Fellow eye) (Eye disorders) | 0 | 1 | 2
ACUTE ELEVATED IOP (Study eye) (Eye disorders) | 2 | 7 | 0
AMD PROGRESSION (Study eye) (Eye disorders) | 6 | 8 | 3
BLEPHARITIS (Study eye) (Eye disorders) | 1 | 0 | 2
CATARACT (Study eye) (Eye disorders) | 8 | 10 | 2
CONJUNCTIVITIS (Study eye) (Eye disorders) | 3 | 0 | 2
DRY EYES (Study eye) (Eye disorders) | 1 | 2 | 4
EYE HEMORRHAGE (Study eye) (Eye disorders) | 5 | 7 | 7
EYE ITCHING (Study eye) (Eye disorders) | 2 | 0 | 0
EYE PAIN (Study eye) (Eye disorders) | 2 | 5 | 2
RETINAL DISORDER (Study eye) (Eye disorders) | 1 | 3 | 1
RETINAL EDEMA (Study eye) (Eye disorders) | 3 | 4 | 0
RETINAL HEMORRHAGE (Study eye) (Eye disorders) | 2 | 2 | 0
RETINAL PIGMENTATION (Study eye) (Eye disorders) | 1 | 1 | 2
SUBRETINAL HEMORRHAGE (Study eye) (Eye disorders) | 3 | 1 | 2
VISION ABNORMAL (Study eye) (Eye disorders) | 4 | 5 | 3
VISION DECREASED (Study eye) (Eye disorders) | 1 | 3 | 3
URINARY TRACT INFECTION (Renal and urinary disorders) | 2 | 5 | 5

LIMITATIONS AND CAVEATS:
Secondary outcome measures were to be assessed at Month 6 and at 24 months. However, this study was not completed but terminated after all patients completed 12 months. Original safety was COSTART now mapped to SOC MedDRA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.